CLINICAL TRIAL: NCT03729024
Title: A Single Center Exploratory Study to Evaluate Uncorrected Distance Vision and Quality of Vision After Light Treatments of an Implanted RxSight Light Adjustable Lens (RXLAL) With The Light Delivery Device (LDD) in Subjects With Preoperative Corneal Astigmatism
Brief Title: Exploratory Study to Evaluate Uncorrected Distance Vision and Quality of Vision After Light Treatments of an Implanted RxSight Light Adjustable Lens (RXLAL) With The Light Delivery Device (LDD) in Subjects With Preoperative Corneal Astigmatism
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: RxSight, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CSP-028
Record Dates: First submitted 2018-10-31; First posted 2018-11-02 (Actual); Results first posted 2021-05-19 (Actual); Last update posted 2021-08-06 (Actual); Status verified 2021-08

CONDITIONS: Aphakia; Cataract
Keywords: Light Adjustable Lens; Intraocular lens; LAL
MeSH Terms: conditions — Aphakia; Cataract

STUDY DESIGN:
Intervention Model Description: All subjects will receive the same treatment; however, each subject will have their eyes randomized to primary or fellow assignment. If only one eye of a patient meets study eligibility, that eye will automatically be designated as the primary eye.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (1):
- Light adjustable lens (LAL) and Light Delivery Device (LDD) (Experimental)
  Interventions: Device: Light Adjustable lens (LAL) and Light Delivery Device (LDD)

INTERVENTIONS:
Device: Light Adjustable lens (LAL) and Light Delivery Device (LDD) — Primary and Fellow eyes will receive Light adjustable lens with Light delivery Device treatments

SUMMARY:
The objective of this study is to evaluate uncorrected distance vision and quality of vision as measured by the McAlinden QoV questionnaire 3 months following the final lock-in treatment of the implanted RxSight Light Adjustable Lens (RxLAL) with the Light Delivery Device (LDD) in subjects with preoperative keratometric astigmatism. This is an exploratory study. No primary effectiveness endpoints will be defined.

ELIGIBILITY:
Inclusion Criteria:

* Must sign a written Informed Consent form and be willing to undergo cataract surgery for unilateral or bilateral implantation of the RxLAL.
* Between the ages of 40 and 80 inclusive on the day the cataract surgery is performed.
* Study eye must have preoperative keratometric cylinder of ≥0.50 D and ≤3.00 D.
* Study eye must have cataract causing reduction in best corrected distance visual acuity (BCDVA) to a level of 20/32 or worse with or without a glare source.
* Willing and able to comply with the requirements for study specific procedures and visits.

Exclusion Criteria:

* Study eye with zonular laxity or dehiscence.
* Study eye with pseudoexfoliation.
* Study eye with age-related macular degeneration involving the presence of geographic atrophy or soft drusen.
* Study eye with diabetes with any evidence of retinopathy.
* Study eye with evidence of glaucomatous optic neuropathy.
* Study eye with history of uveitis.
* Study eye with prior history of Intacs, Radial keratotomy (RK), Conductive keratoplasty (CK), Astigmatic keratotomy (AK), Phakic Implantable Collamer Lens (ICL), Corneal Inlay, or with previous pterygium excision unless the pterygium did not extend more than 2mm onto the cornea from the limbus.
* Subjects taking systemic medication that may increase sensitivity to UV light.
* Subjects taking a systemic medication that is considered toxic to the retina such as tamoxifen.
* Study eye with history of ocular herpes simplex virus.
* Study eye with history of a congenital color vision defect

Ages: 40 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 21 (Actual)
Dates: Start 2018-01-26 (Actual); Primary Completion 2019-04-15 (Actual); Study Completion 2020-02-04 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- CODET Vision Institute, Tijuana, Mexico

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Units Other Than Participants: Eyes
Period: Overall Study
Arm/Group | Light Adjustable Lens (LAL) and Light Delivery Device (LDD)
Started | 21; 42 Eyes
Completed | 21; 42 Eyes
Not Completed | 0; 0 Eyes

BASELINE CHARACTERISTICS:
Units Other Than Participants: Eyes
Arm/Group | Light Adjustable Lens (LAL) and Light Delivery Device (LDD)
Number analyzed (Participants) | 21
Number analyzed (Eyes) | 42
Age, Continuous [Mean (Standard Deviation); unit: years] | 68.3 (5.3)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 12
  Male | 9
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 18
  Not Hispanic or Latino | 3
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  Mexico | 21

OUTCOME MEASURES:

1. Primary Outcome: Percent of Eyes With UCDVA of 20/20 or Better
Time Frame: 6 months
Measure: Count of Units; unit: Eyes
Units Other Than Participants: Eyes
Arm/Group | Light Adjustable Lens (LAL) and Light Delivery Device (LDD)
Number analyzed (Participants) | 21
Number analyzed (Eyes) | 42
Eyes | 41

ADVERSE EVENTS:
Time Frame: Through study completion, an average of 6 months
Description: The at Risk number in All-Cause Mortality represent whole participants while the at Risk number in the Serious and Other (Not Including Serious) Adverse Events tables represent the number of eyes. Non-ocular adverse events were not collected.
Arm/Group | Light Adjustable Lens (LAL) and Light Delivery Device (LDD)
All-Cause Mortality (participants affected / at risk) | 0/21
Serious Adverse Events (participants affected / at risk) | 0/42
Other Adverse Events (participants affected / at risk) | 1/42
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Light Adjustable Lens (LAL) and Light Delivery Device (LDD) (N=42)
Cystoid Macular Edema (Eye disorders) | 1 (1) — Corneal Edema (corneal swelling (stromal or epithelial) resulting in BCDVA ≤ 20/40 after Postop Week 3

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2018-04-27): https://cdn.clinicaltrials.gov/large-docs/24/NCT03729024/Prot_SAP_000.pdf